CLINICAL TRIAL: NCT03269578
Title: Longitudinal Sample Collection and Tracking for the Developmental Therapeutics Clinic, National Cancer Institute
Brief Title: Sample Collection and Tracking for the Developmental Therapeutics Clinic
Status: Recruiting | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 170156; 17-C-0156
Record Dates: First submitted 2017-08-31; First posted 2017-09-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06-27

CONDITIONS: Neoplasms; Lymphoma
Keywords: Pharmacodynamics; Tissue Collection; Tissue Biopsies; Biospecimen; Assay Development; Natural History
MeSH Terms: conditions — Neoplasms; Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 1: Patients with cancer or benign tumors being treated on NCI/DTC studies

SUMMARY:
Background:

People who join a study in the Developmental Therapeutics Clinic (DTC) have tests. These include blood draws and biopsies. Researchers collect data from these samples. Some people take part in more than one study at the DTC. At this time, data are connected only with one single study. Researchers want to access people s medical records. This will allow them to link the research data from all their studies they have or will take part in. Researchers also want to collect medical data about their diagnosis and treatment history. This will allow them to see how their cancer reacted to different drugs over time.

Objective:

To enter people into a master protocol to connect research sample and treatment data across DTC studies.

Eligibility:

People ages 18 and older who are being evaluated or treated for cancer in the DTC

Design:

Participants will allow researchers to look at all the data from their research samples. This includes those from their current, past, and any future NIH studies.

Participants will allow researchers to access some of their medical data. This includes age, diagnosis, treatment history, and response to treatment.

Participants will provide no new samples.

...

DETAILED DESCRIPTION:
Background:

Research samples and data collected on a treatment-intent protocol are discrete items associated with that protocol up until the patient comes off study, usually due to disease progression. These data are not stored in the patient s medical records, but are essential to understand tumor response to different drugs over time. Patients in the Developmental Therapeutics Clinic (DTC) often start other clinical trials; this protocol provides a mechanism to connect research data about that patient from one trial to the next as long as the patient remains eligible and has given his or her informed consent. No new analysis will be performed under this protocol.

There is research interest in collecting pre- and post-dose research biopsies and other samples such as circulating tumor cells to measure dynamic drug-specific target effects (e.g., changes in epithelial-mesenchymal transition, DNA damage response, or immunotherapeutic cell infiltration), and then to evaluate molecular changes before and during disease progression to understand why the tumors initially respond but then became resistant to treatment.

To accomplish this, we will connect research results from consecutive trials with limited patient information (age, sex, disease, prior therapies, protocol number/drug regimen, response, and duration of treatment).

Each patient who consents to participate in this non-treatment, longitudinal sample protocol agrees to allow his or her Medical Record Number (MRN) to be used to track participation on DTC clinical trials.

Objectives:

Patients will be entered onto this "master" longitudinal protocol to connect research sample and treatment data across consecutive DTC clinical trials.

Biopsy samples collected at time of disease progression on one research trial will be evaluated for use as the baseline sample for the next research trial, potentially obviating the need for additional biopsies.

Eligibility:

Adult patients who are being evaluated for and/or treated for cancer or benign tumors at the DTC.

Design:

No samples will be collected under this longitudinal protocol, no treatment decisions will be made based on data collected, and no new analysis will be performed.

Specimens for research purposes, as outlined in this protocol, will be those obtained from tests and procedures that are done as required by the primary research protocols that a given patient is enrolled in. Tissue collected under DTC tissue procurement protocol 06-C-0213 will not be used or tracked.

Sample location and use will be managed in the Repository at the Frederick National Laboratory for Cancer Research using LabMatrix software.

Patients may remain on this longitudinal protocol for the duration of their consent.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Patients who are being evaluated and/or treated for cancer or benign tuumors in the Developmental Therapeutics Clinic at the NIH Clinical Center
* Ability to understand and willingness to sign a written informed consent document indicating their willingness to have data from their tissue or biologic fluid research specimens and limited medial information used for research as outlined in this protocol and to allow protocol staff access to the CRIS database and their Medical Records Number (MRN).
* Age greater than or equal to 18 years

ECLUSION CRITERIA:

None

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients on research protocols at the Developmental Therapeutics Clinic
Sampling Method: Non-Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2017-08-28 (Actual); Primary Completion 2027-05-23 (Estimated); Study Completion 2027-05-30 (Estimated)

PRIMARY OUTCOMES:
Obtaining informed consent | Time of enrollment
  Collation of research sample and treatment data from individual patients across their participation in consecutive DTC clinical trials

CONTACTS AND LOCATIONS:
Overall Officials: Alice P Chen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2017-C-0156.html